CLINICAL TRIAL: NCT02660632
Title: Effect of Thoracic Epidural Analgesia vs Rectus Sheath Catheters on Postoperative Pulmonary Function After Midline Laparotomy: A Prospective Randomized Controlled Study
Brief Title: Epidural Block vs. Rectus Sheath Block on Postoperative Pulmonary Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R ∕ 15.12.48
Record Dates: First submitted 2016-01-16; First posted 2016-01-21 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Abdominal Surgeries
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thoracic epidural analgesia (TEA) (Placebo Comparator): Patients who will be subjected for midline laparotomy, will receive epidural analgesia through an inserted thoracic epidural catheter before induction of general anesthesia
  Interventions: Other: Thoracic epidural analgesia (TEA)
- Rectus sheath catheter block (Active Comparator): After insertion of bilateral rectus sheath catheters, 20 ml of 0.25% bupivacaine will be injected on each side, then continuous infusion pumps will be connected to the catheters and set to deliver boluses of 20 mL of 0.25% bupivacaine, with a 4-hour lockout for up to 48 h postoperatively.
  Interventions: Other: Rectus sheath catheter block

INTERVENTIONS:
Other: Thoracic epidural analgesia (TEA) — Epidural catheter will be inserted at T9-T11. Then, epidural analgesia will be activated with administering bolus of 10 mls 0.25% bupivacaine in conjunction with100 mcg fentanyl to establish a block. This will be followed by an infusion of 0.125% bupivacaine in conjunction with 2 mcg/ ml fentanyl at a rate of 10 mls /hour and then titrated to effect for up to 48 hour postoperative
  Arms: Thoracic epidural analgesia (TEA)
Other: Rectus sheath catheter block — Following insertion of bilateral rectus sheath catheters, 20 ml of 0.25% bupivacaine will be injected through each one. Then continuous infusion pumps will be connected to the catheters and set to deliver boluses of 20 mL of 0.25% bupivacaine, with a 4-hour lockout for up to 48 h postoperatively.
  Arms: Rectus sheath catheter block

SUMMARY:
Pulmonary complications are among the most important postoperative complications after midline incisions, for which different analgesic modalities have been tried.

Epidural analgesia is the recommended technique to relieve pain after major abdominal surgery owing to the proved superior analgesia, reduction of opioid related side effects as nausea, vomiting, pruritis and sedation, earlier recovery of bowel function and earlier ability for postoperative mobility However, it is not without complications.

Rectus sheath block provides several advantages over epidural anesthesia. It lessens the potential risks associated with neuraxial techniques, so it may represent a novel alternative approach for somatic analgesia after major abdominal surgeries. Although patients with rectus sheath block may experience some visceral pain, it is usually minimal by 24 hours after surgery.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of thoracic epidural analgesia and rectus sheath blockade on postoperative pulmonary functions, pain scores, duration of analgesia, sedation scores, patients' satisfaction and adverse effects.

FEV1, FEV1/FVC ratio will be measured by a bed side spirometer.

* Induction of anesthesia: propofol 1.5-2.5 mg kg-1.
* Muscle Relaxants: rocuronium 0.6 mg kg-1 for induction.
* Maintenance: Sevoflurane 0.7-1.5 MAC vaporized in air-oxygen (40% inspired fraction).

Radial artery catheterization: under complete aseptic conditions 20G cannula will be inserted into the radial artery of non-dominant hand after performing modified Allen's test and local infiltration of 0.5ml xylocaine 2% .

Thoracic epidural catheter will be inserted before induction of general anaesthesia under aseptic insertion conditions and using loss of resistance to air technique with the patient in the sitting position at T9- T11 interspaces.

The Rectus sheath catheters will be inserted bilaterally using ultrasound (SonoSite M-Turbo®, Sonosite , USA) guidance as described by Webster after induction of general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class I to III.
* Patients scheduled for elective midline laparotomy.

Exclusion Criteria:

* Morbid obese patients.
* Severe or uncompensated cardiovascular disease.
* Significant renal disease.
* Significant hepatic disease.
* Pregnancy.
* Lactating.
* Allergy to the study medications.
* Psychological disorder.
* Neurological disorder.
* Communication barrier.
* Mental disorders.
* Epilepsy.
* FEV1 or FEV1/FVC ratio less than 50%, dyspnea with a New York Heart Association class IV.
* Drug or alcohol abuse.
* Contraindications to epidural anaesthesia.
* Opioid analgesic medication within 24 h before the operation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Changes in forced expiratory volume in 1 second (FEV1) | Before and for 72 hours after surgery
Changes in ratio between forced expiratory volume in 1 s and forced vital capacity (FEV1/FVC) | Before and for 72 hours after surgery

SECONDARY OUTCOMES:
Changes in arterial blood gases | Before and for 72 hours after surgery
Visual analog pain scores | for 48 hours after surgery
  Postoperative pain will be assessed on rest and with cough and during movements for both of visceral and parietal pain
Sedation score | for 48 hours after surgery
  Sedation scores using a sedation scale (awake and alert= 0; quietly awake= 1; asleep but easily roused= 2; deep sleep= 3.
Postoperative nausea and vomiting | for 48 hours after surgery
  The degree of nausea and vomiting. Nausea will be measured using a numerical rating system (none= 0; mild= 1; moderate= 2; severe= 3). The number of vomiting episodes and the number of anti-emetics received
Return of bowel function | for 72 hours after surgery
  The times to first flatus, defecation, intake of clear liquid and solid food tolerance
Time to hospital discharge | for 15 days after surgery
  from the end of anesthesia
Cumulative tramadol use | For 48 hours after surgery
Overall patient's satisfaction | For 48 hours after surgery
  Patient overall satisfaction will be assessed before hospital discharge using the visual analog score
Intraoperative use of ephedrine | For 5 hours after induction of anesthesia
Postoperative cardio-respiratory complications | For 7 days after surgery
Postoperative wound infection | For 21 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Samah Elkenany, MD, Principal Investigator — Lecturer of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura university, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided